CLINICAL TRIAL: NCT03546231
Title: Clinical and Echocardiographic Characteristics and Prognosis of trIcuspid regurgiTation (EPIT): Prospective and Retrospective Follow-up of a Cohort of Patients With Moderate or Severe Tricuspid Regurgitation
Brief Title: Characteristics and Prognosis of Moderate or Severe Tricuspid Regurgitation
Acronym: EPIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0027
Record Dates: First submitted 2018-04-13; First posted 2018-06-06 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Tricuspid Valve Disease
Keywords: Tricuspid regurgitation; tricuspid valve; surgery; outcome; prognosis; mortality; right ventricle; asymptomatic
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The tricuspid valve : its evaluation is relatively difficult in echocardiography and the management of tricuspid valve diseases remains poorly codified.

DETAILED DESCRIPTION:
The tricuspid valve is often called the "forgotten valve" because its evaluation is relatively difficult in echocardiography and the management of tricuspid valve diseases remains poorly codified. In developed countries, TR is mainly functional, related to a remodeling of the right cavities in response to an increase in the load conditions. This remodeling induces a dilation of the tricuspid ring and / or a "tenting" of the tricuspid leaflets. Once TR is present, a vicious circle settles because TR increases right ventricle dilation. Transthoracic echocardiography is the key examination allowing noninvasive, quantification and assessment of hemodynamic repercussions of TR.

TR remains asymptomatic for a long time, often diagnosed with a significant delay at the stage of advanced right heart failure. At this stage, the surgical risk is important, at least more important than for left heart valve diseases and it is therefore essential to define the right time for proposing valvular surgery to patients. Indeed, TR is an independent factor of mortality and only surgical treatment improves the prognosis.

Current guidelines remain vague given the low number of prognostic studies and of their contradictory results often influenced by the significant comorbidities of patients, the presence of pulmonary hypertension or left heart valve disease. Only a minority of patients (<1%) is referred to surgery because operative mortality is often judged unacceptable in elderly patients or in cases of advanced right ventricular dysfunction.

The constitution of a prospective and retrospective cohort will improve the state of knowledge on etiologies, natural history, prognosis and management of patients with moderate or severe TR.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 ans
* inclusion criteria: moderate or severe tricuspid regurgitation
* exclusion criteria: Refusal to participate/ prior surgery of the tricuspid valve

Min Age: 18 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate or severe tricuspid regurgitation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 Years
  It corresponds to the delay between the diagnostic and the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe TRIBOUILLOY, Pr, Principal Investigator — CHU AMIENS-PICARDIE
Locations (1):
- CHU Amiens-Picardie, Amiens, France